CLINICAL TRIAL: NCT06832423
Title: CAN CREATINE SUPPLEMENTATION IMPROVE PERFORMANCE in ROCK CLIMBERS?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain dietary intervention due to manufacturer withdrawing product from market.
Sponsor: Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: creatine01; 15/WA/0438 (Other: Wales Research Ethics Committee 5)
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Rock Climbing
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Creatine (Experimental): 5g of the active supplement (creatine monohydrate) will be consumed four times per day for five days (the "loading phase"). Thereafter the dose will be reduced to 3 g once per day for twelve weeks (the "maintenance phase").
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): 5g of the placebo supplement (fructose supplement providing the same calorie content as the creatine) will be consumed four times per day for five days (the "loading phase"). Thereafter the dose will be reduced to 3 g once per day for twelve weeks (the "maintenance phase").
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Powder mixed with flavoured water
  Arms: Creatine
Dietary Supplement: Placebo — Powder mixed with flavoured water
  Arms: Placebo

SUMMARY:
Why? Bouldering is a form of rock climbing that comprises short rock climbs of approximately three metres in height. Approximately 35,000 people participate in bouldering the UK, 200 of whom do so competitively. Bouldering requires a high strength to body weight ratio. Creatine is widely used in other sports as a nutritional supplement to increase muscle mass, strength and exercise tolerance. Whether Creatine can enhance performance of elite boulderers and in other disciplines of climbing is not known. Answering this question is important to identify safe and legal performance enhancing aids to enable recreational and competitive boulderers and climbers to maximise their personal and competitive potential.

What? This study will investigate a nutritional supplement, Creatine monohydrate (the "active supplement"), and compare its efficacy to a nondistinguishable and similar calorie content supplement, fructose (the "placebo"). Who? Elite boulderers from the Great Britain (GB) Bouldering Team will be invited to take part. If recruitment is slow, highly accomplished climbers from the North Wales region will also be invited.

Where? The study data collection visits will be completed at Bangor University. The supplementation will be completed by the participants at home.

How? The study will utilise a randomised placebo controlled trial design. Randomised means that participants will be allocated to receive the active supplement OR the placebo by chance. The study will last 18 weeks. Participants will visit the University for familiarisation (week 4) and again at baseline (week 0). The tests will include assessment of body weight, a whole body xray scan to determine skeletal muscle mass (at week 0 and 13 only), tests of upper body and core muscle strength, and a test of climbing-specific performance during a simulated bouldering competition.

Then, depending on group allocation, 5 g of the active supplement or placebo will be consumed four times per day for five days (the "loading phase"). Thereafter the dose will be reduced to 3 g once per day for twelve weeks (the "maintenance phase"). The supplement and the placebo will be mixed with flavoured water and consumed at meal and snack times.

Finally, at study cessation (week 13), the University visit will be repeated. The research is being funded by Bangor University. The creatinine and placebo supplements are being supplied by a nutritional company that has no influence over the publication of the results.

ELIGIBILITY:
Inclusion Criteria:

* membership of the GB Bouldering Team or climbing at grade above F6c

Exclusion Criteria:

* evident or previously diagnosed kidney damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
ALM | 12 weeks
  Appendicular lean mass change (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Bangor University, Bangor, Gwynedd, United Kingdom

IPD SHARING:
Plan to Share IPD: No